CLINICAL TRIAL: NCT07379073
Title: Evaluation of a Clinical Support Website for the Management of Common Mental Health Conditions in Primary Care on Compliance With Benzodiazepine Prescribing Recommendations
Acronym: Psycho-MG
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: MSPU de Pins-Justaret (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Psycho-MG
Record Dates: First submitted 2026-01-23; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Benzodiazepine Use

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (trained on PsychoMG website) (Experimental): Training intervention on benzodiazepine prescribing with access to the PsychoMG website providing evidence-based clinical decision algorithms for anxiety and sleep disorder management.
  Interventions: Other: Training
- Control Group (No Intervention): Training intervention on benzodiazepine prescribing without access to the PsychoMG website providing evidence-based clinical decision algorithms for anxiety and sleep disorder management.

INTERVENTIONS:
Other: Training — Training intervention on benzodiazepine prescribing with access to the PsychoMG website providing evidence-based clinical decision algorithms for anxiety and sleep disorder management.
  Arms: Experimental Group (trained on PsychoMG website)

SUMMARY:
This cluster-randomized study aims to evaluate the impact of a web-based clinical support tool on adherence to recommended maximum durations for benzodiazepine prescriptions among new users in primary care. General practitioners (GPs) participating in the study will have access to the website, which provides evidence-based algorithms for the management of common mental health conditions, including anxiety and sleep disorders. Prescription data and patient characteristics will be extracted from the French national health insurance database (DCIR). The primary outcome is the proportion of new benzodiazepine users whose prescriptions comply with recommended duration guidelines. Multilevel logistic regression models will assess the intervention effect, adjusting for patient- and GP-level factors.

ELIGIBILITY:
Inclusion criteria:

* Being a general practitioner or a specialist in general medicine.
* Practicing in the Occitanie region.
* Working in private practice.
* Being registered under Sector 1 fee agreements.
* Providing informed consent to participate in the study.
* Having computer equipment in the medical office, available during consultation (desktop, laptop, tablet, or smartphone) with internet access.

Exclusion criteria:

- Physicians who have been practicing for less than two years, as they are unlikely to have sufficient retrospective data on prescription reimbursements for their patients.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2027-10-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
Compliance with recommended maximum duration of benzodiazepine prescriptions among new users | 12 months
  Primary outcome measure: adherence to recommended prescription duration (yes/no) for benzodiazepines
  A patient is considered to have a prescription duration for benzodiazepines that is either adherent or non-adherent if they had no benzodiazepine exposure in the previous year and their duration of exposure during the first treatment episode:
  1. is less than 12 weeks for anxiolytic benzodiazepines,
  2. is less than 28 days for hypnotic benzodiazepines and related drugs, in accordance with current recommendations.